CLINICAL TRIAL: NCT05407922
Title: Laparoscopic Value in the Management of Acute Abdomen During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Emad Ali Ahmed Ali, Lecturer, Sohag University
Other Study IDs: soh-med-42342
Record Dates: First submitted 2022-05-27; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Acute Abdomen; Pregnancy Related
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopy Group: The laparoscopy group included every pregnant woman having laparoscopic intervention because of acute abdominal pain during any trimester of her pregnancy.
  Interventions: Procedure: Laparoscopy vs Non-laparoscopy approach
- Non-laparoscopy Group: Non-laparoscopy Group included every pregnant woman having treatment approach other than the laparoscopic approach because of acute abdominal pain.
  Interventions: Procedure: Laparoscopy vs Non-laparoscopy approach

INTERVENTIONS:
Procedure: Laparoscopy vs Non-laparoscopy approach — Pregnant women who will undergo a laparoscopic or open surgical exploration of the abdomen

SUMMARY:
The term "acute abdomen" is often used to describe the manifestations of any serious intraperitoneal disease, which may indicates surgical intervention. Acute abdomen in pregnancy accounts for approximately 7-10% of all abdominal emergencies.

Several pathologies could contribute acute abdominal pain during pregnancy. They include obstetric and non-obstetric causes. As for the non-obstetric causes , any gastrointestinal or urological disorders could be presented by an acute abdominal pain.

In pregnancy, several factors overlap and making the diagnosis challenging. These factors include the distorted anatomy by the growing uterus that displaces intraperitoneal structures. Additionally, nausea, vomiting, and abdominal pain are considered the normal course during pregnancy especially at the first trimester. Moreover, sure diagnosis must be achieved to operate in a pregnant woman with more possible morbidity and mortality for the mother and\or fetus.

DETAILED DESCRIPTION:
Laparoscopy can be safely performed during any trimester of pregnancy. Historical recommendations were to limit surgery to the second trimester only, but these recommendations were based on experience with open surgical procedures during pregnancy. These recommendations were thought to minimize the spontaneous abortion rate of surgical intervention during the first trimester, which was reported to be as high as 12%, and to avoid preterm labor, reported in up to 40%, when surgery occurred during the third trimester. However, studies limited to laparoscopy have shown improved outcomes and demonstrated that pregnant patients may undergo laparoscopic surgery safely during any trimester without any appreciated increase in risk to the mother or fetus.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women having acute abdomen and underwent surgical intervention will be included in this study.

Exclusion Criteria:

* Non-pregnant women with acute abdomen are excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant females
Study Population: Any pregnant woman presented with acute abdominal pain to the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Early complications for the mother and fetus | through study completion, an average of 1 year
  during the postoperative hospital stay

SECONDARY OUTCOMES:
Late complications for the mother and fetus | 30 days
  during the first 30 days postoperatively

IPD SHARING:
Plan to Share IPD: Undecided
may be all data but after publication

REFERENCES:
- [Background] Augustin G, Majerovic M. Non-obstetrical acute abdomen during pregnancy. Eur J Obstet Gynecol Reprod Biol. 2007 Mar;131(1):4-12. doi: 10.1016/j.ejogrb.2006.07.052. Epub 2006 Sep 18. PMID 16982130
- [Background] Di Saverio S, Podda M, De Simone B, Ceresoli M, Augustin G, Gori A, Boermeester M, Sartelli M, Coccolini F, Tarasconi A, De' Angelis N, Weber DG, Tolonen M, Birindelli A, Biffl W, Moore EE, Kelly M, Soreide K, Kashuk J, Ten Broek R, Gomes CA, Sugrue M, Davies RJ, Damaskos D, Leppaniemi A, Kirkpatrick A, Peitzman AB, Fraga GP, Maier RV, Coimbra R, Chiarugi M, Sganga G, Pisanu A, De' Angelis GL, Tan E, Van Goor H, Pata F, Di Carlo I, Chiara O, Litvin A, Campanile FC, Sakakushev B, Tomadze G, Demetrashvili Z, Latifi R, Abu-Zidan F, Romeo O, Segovia-Lohse H, Baiocchi G, Costa D, Rizoli S, Balogh ZJ, Bendinelli C, Scalea T, Ivatury R, Velmahos G, Andersson R, Kluger Y, Ansaloni L, Catena F. Diagnosis and treatment of acute appendicitis: 2020 update of the WSES Jerusalem guidelines. World J Emerg Surg. 2020 Apr 15;15(1):27. doi: 10.1186/s13017-020-00306-3. PMID 32295644
- [Background] Zachariah SK, Fenn M, Jacob K, Arthungal SA, Zachariah SA. Management of acute abdomen in pregnancy: current perspectives. Int J Womens Health. 2019 Feb 8;11:119-134. doi: 10.2147/IJWH.S151501. eCollection 2019. PMID 30804686
- [Background] Jackson H, Granger S, Price R, Rollins M, Earle D, Richardson W, Fanelli R. Diagnosis and laparoscopic treatment of surgical diseases during pregnancy: an evidence-based review. Surg Endosc. 2008 Sep;22(9):1917-27. doi: 10.1007/s00464-008-9989-6. Epub 2008 Jun 14. PMID 18553201